CLINICAL TRIAL: NCT03096808
Title: A Prospective Non-Inferiority Trial of the Use of Adaptive Radiotherapy for Head and Neck Cancer Undergoing Radiation Therapy
Brief Title: Adaptive Radiotherapy for Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-148
Record Dates: First submitted 2017-03-15; First posted 2017-03-30 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Head and Neck Cancer; Paranasal Sinus Cancer; Oropharynx Cancer; Oral Cavity Cancer; Nasopharynx Cancer; Larynx Cancer; Hypopharynx Cancer
Keywords: adaptive radiotherapy; ART; intensity modulated radiation therapy; IMRT
MeSH Terms: conditions — Head and Neck Neoplasms; Paranasal Sinus Neoplasms; Oropharyngeal Neoplasms; Mouth Neoplasms; Nasopharyngeal Neoplasms; Laryngeal Neoplasms; Hypopharyngeal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adaptive Radiotherapy (Experimental): Eligible patients will receive IMRT of 60-70Gy in 30-35 once-daily fractions with or without concurrent chemotherapy according to the current standard of care.
  Interventions: Radiation: Adaptive Radiotherapy

INTERVENTIONS:
Radiation: Adaptive Radiotherapy — ART involved modification of the radiation treatment plan during treatment course to account for temporal variations in anatomy due to changes in tumor volume and/or patients' weight loss.
  Other Names: ART

SUMMARY:
The purpose of this study is to demonstrate that adaptive radiotherapy (ART) in head and neck cancer patients are comparable to historical controls in head and neck patients undergoing standard intensity-modulated radiation therapy (IMRT) without ART.

ELIGIBILITY:
Inclusion Criteria:

* Participants with pathologically confirmed cancers of paranasal sinuses, oropharynx, oral cavity, nasopharynx, larynx, hypopharynx, and unknown primary and will receive definitive radiation therapy with or without chemotherapy.
* Karnofsky performance status >= 70%
* Women of childbearing potential need to have a negative serum pregnancy test at the time of therapy
* Participants must have the ability to understand and the willingness to sign a written consent form

Exclusion Criteria:

* Female participants who are pregnant or breast feeding
* Participants who are not able to comply with study and/or follow up procedures
* Participants who have received induction chemotherapy before radiation treatment
* Participants who had prior head and neck radiation therapy
* Participants who are enrolled in a national/international cooperative group trials
* Patients with metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2021-10-22 (Actual)

PRIMARY OUTCOMES:
Number of patients with locoregional recurrence-free interval | 2 years
  This is assessed by imaging studies and/or physical exams at follow- up visits. This will include a diagnostic FDG PET/CT scan. CT and/or MRI of the primary site and neck will also be recommended. Patients will be classified as locoregional recurrence-free as long as there is no evidence of locoregional recurrence of disease by clinical evaluation, CT, MRI, and/or PET-CT according to the standard of care. For patients achieving complete response of disease, no further imaging study is necessary.

CONTACTS AND LOCATIONS:
Overall Officials: C. Jillian Tsai, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memoral Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org